CLINICAL TRIAL: NCT02868970
Title: Pharmacists as Immunizers to Improve Coverage and Provider/Recipient Satisfaction: A Prospective, Controlled Community Embedded Study With Vaccines With Low Coverage Rates (The Improve ACCESS Study)
Brief Title: Pharmacists as Immunizers to Improve Coverage and Provider/Recipient Satisfaction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Canadian Immunization Research Network (Network)
Collaborators: GlaxoSmithKline (Industry); MCM Vaccines B.V. (Industry); Canadian Center for Vaccinology (Other); Dalhousie University (Other)
Responsible Party: Principal Investigator, Jennifer Isenor, Principal Investigator, Canadian Immunization Research Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CT12
Record Dates: First submitted 2016-07-11; First posted 2016-08-16 (Estimated); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Healthy
MeSH Terms: interventions — 4CMenB vaccine; Influenza Vaccines; Herpes Zoster Vaccine; Hepatitis A Vaccines; Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community (2 in NB, 2 from NS) (Other): There are four communities involved in the study, two in New Brunswick and two in Nova Scotia. All pharmacies in each community will be allocated to one intervention. Interventions include: High-Dose TIV, Meningococcal B Vaccine, Meningococcal ACWY vaccine, Tdap, Herpes Zoster vaccine and Travel Health vaccines (Hepatitis A, Hepatitis B, Typhoid Fever).
  Interventions: Biological: Meningococcal B; Biological: High-Dose TIV; Biological: Tdap (tetanus-diphtheria-acellular pertussis); Biological: Meningococcal ACWY; Biological: Herpes Zoster; Biological: Travel Health (Hepatitis A, Hepatitis B, Typhoid Fever)

INTERVENTIONS:
Biological: Meningococcal B — Bexsero is indicated for active immunisation of individuals from 2 months of age and older against invasive meningococcal disease caused by Neisseria meningitidis group B.
  Other Names: Bexsero
Biological: High-Dose TIV — Fluzone High-Dose is an injectable influenza vaccine made to protect against the flu strains most likely to cause illness for that particular flu season.
  Other Names: FluZone
Biological: Tdap (tetanus-diphtheria-acellular pertussis) — Tdap is a combination vaccine that protects against three potentially life-threatening bacterial diseases: tetanus, diphtheria, and pertussis (whooping cough).
Biological: Meningococcal ACWY — Meningococcal ACWY vaccine is indicated for active immunization of individuals up to 55 years of age against invasive meningococcal diseases caused by Neisseria meningitides serogroups A, C, W-135 and Y.
Biological: Herpes Zoster — Herpes zoster vaccine is indicated for the immunization of individuals 50 years of age or older for the prevention of herpes zoster (shingles).
Biological: Travel Health (Hepatitis A, Hepatitis B, Typhoid Fever) — Hepatitis A vaccine is indicated for immunization against infections caused by hepatitis A virus; Hepatitis B vaccine is indicated for immunization against infection caused by hepatitis B virus; and typhoid fever vaccine is indicated for active immunization against Salmonella typhi, the organism which causes typhoid fever.

SUMMARY:
This project proposes to implement and compare new community pharmacy-based strategies for improving vaccine coverage.

DETAILED DESCRIPTION:
Although there are many safe and effective vaccines for adults, the Public Health Agency of Canada has noted that public perception of vaccination is that it is primarily for infants and children. The National Advisory Committee on Immunization (NACI) recommends adults and adolescents receive the influenza vaccine, tetanus-diphtheria-acellular pertussis vaccine (Tdap), and meningococcal vaccines (MenACWY, 4CMenB). As well, NACI recommends that people 60 years or older receive the herpes zoster vaccine and that Canadians who travel to high-risk areas should consider getting vaccinated to protect themselves against travel-related illnesses, such as Hepatitis A and Typhoid Fever. While NACI makes recommendations, provinces and territories (P/Ts) determine if they will fund and implement vaccine programs. Unlike the childhood immunization programs which tend to be funded by P/Ts, many adult vaccines are unfunded, resulting in poor population uptake. In this project,the investigators propose to implement and compare new community pharmacy-based strategies for improving vaccine coverage.

Patients are typically educated about preventative health care during face-to-face visits with physicians in office settings. The ability to educate and deliver preventative health care is limited by the available provider time during office visits - providers often focus on acute needs and current disease management. New delivery models and a means of extending preventative health care delivery outside of traditional face-to-face office visits are needed.

Pharmacists are in a unique position of being among the most accessible of health professionals. Given their extended operating hours, accessibility, and established trust with patients, pharmacists are well-positioned to improve vaccination rates and health system efficacy through injection administration.

Vaccine coverage rates will be measured using the following:

1. pharmacy database analysis,
2. public health vaccine reports by physicians,
3. number of vaccine doses delivered to pharmacies in all four regions, and
4. public survey within the study communities to determine immunization status.

Intervention communities include Saint John, New Brunswick and New Glasgow/Pictou/Antigonish, Nova Scotia area, which include the smaller towns of Stellarton and Westville, Nova Scotia. Control communities include Moncton, New Brunswick and Kentville/New Minas/Wolfville, Nova Scotia, which include the smaller towns of Canning and Coldbrook, Nova Scotia.

ELIGIBILITY:
Inclusion criteria:

* For the selection of the four communities include population size (approximately 30,000 adults >18 years of age), stable population, service by a centralized regional hospital and local community hospitals, availability of community pharmacies, interest of community pharmacists (sufficient numbers of pharmacists qualified to provide vaccinations), and lack of substantial health care spill over to adjacent communities.
* Spill over is defined as a pattern of health-care utilization where patients regularly receive care at different regional health centers.
* Intervention communities include Saint John, New Brunswick and New Glasgow/Pictou/Antigonish, Nova Scotia area, which include the smaller towns of Stellarton and Westville, Nova Scotia.
* Control communities include Moncton, New Brunswick and Kentville/New Minas/Wolfville, Nova Scotia, which include the smaller towns of Canning and Coldbrook, Nova Scotia.

Exclusion criteria: Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2404 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott A Halperin, MD, Principal Investigator — Dalhousie
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pharmacies were recruited from four communities in Nova Scotia and New Brunswick, Canada. One community in each province served as the intervention community, where community pharmacies were allocated to implement various strategies designed for each of the target vaccines. One community in each province also served as the non-intervention community, where immunization practice continued unchanged. Intervention and non-intervention pharmacies were assigned to each group rather than participants.
Units Other Than Participants: Pharmacies
Groups:
- Intervention Communities: One community in each Nova Scotia and New Brunswick served as the intervention site where pharmacists in the community pharmacies were allocated to implement various strategies specifically designed for each of the target vaccines (tetanus-diphtheria-acellular pertussis (Tdap), high-dose influenza (HD flu), meningococcal B (4CMenB), meningococcal ACWY (MenACWY), travel health (hepatitis A & B, typhoid fever), and herpes zoster vaccines). The pharmacists applied various strategies, which included: combining vaccinations with other services such as influenza vaccine seasonal campaigns, back to school pharmacy services, travel season and standard services; targeted patient outreach; promotion of immunization weeks; and social media messaging, signage, handouts, and bag stuffers to promote the study vaccines. Intervention pharmacies were provided with support materials and received background information and training about the vaccines through in-person and/or web-based video conferences.
- Non-Intervention Communities: One community in each Nova Scotia and New Brunswick served as the non-intervention site where immunization practice continued unchanged, and pharmacists would administer vaccines when requested or when deemed appropriate during routine care. Pharmacies in non-intervention communities continued their standard immunization practices without any study-related education, training, or outreach.
Period: Overall Study
Arm/Group | Intervention Communities | Non-Intervention Communities
Started | NA; 23 Pharmacies (Information on the number of participants is not available (NA) because no participants were assigned to this arm/group. Instead, pharmacies from the selected community in each province were assigned to the "Intervention Communities" arm/group.) | NA; 25 Pharmacies (Information on the number of participants is not available (NA) because no participants were assigned to this arm/group. Instead, pharmacies from the selected community in each province were assigned to the "Non-Intervention Communities" arm/group)
Completed | NA; 23 Pharmacies (Information on the number of participants is not available (NA) because no participants were assigned to this arm/group. Instead, pharmacies from the selected community in each province were assigned to the "Intervention Communities" arm/group.) | NA; 21 Pharmacies (Information on the number of participants is not available (NA) because no participants were assigned to this arm/group. Instead, pharmacies from the selected community in each province were assigned to the "Non-Intervention Communities" arm/group)
Not Completed | NA; 0 Pharmacies | NA; 4 Pharmacies

BASELINE CHARACTERISTICS:
Population: Information on the number of participants is not available (NA) because no participants were assigned to the arms/groups. Instead, pharmacies from the selected community in each province were assigned to each arm/group. Pharmacies were not assessed for these baseline measures; therefore, data were not collected and cannot be reported.
Units Other Than Participants: Pharmacies
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Communities | Non-Intervention Communities | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Pharmacies) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Number of Vaccines Administered by Participating Pharmacies in the Intervention and Non-intervention Communities Before and During the Intervention.
Description: A 2-year demonstration program was conducted in two Canadian provinces (New Brunswick and Nova Scotia). One community in each province served as the intervention community, where pharmacies were allocated to implement various strategies specifically designed for each of the target vaccines. One community in each province also served as the non-intervention community, where immunization practice continued unchanged. Vaccine uptake was compared using pharmacy-generated reports of the number of vaccine doses administered before (from September 2015 to August 2017) and during (September 2017 to November 2019) the intervention and between non-intervention and intervention pharmacies.
Time Frame: At the time of vaccination, 1 day over two years from September 2017 to November 2019.
Population: Information on the number of participants is not available (NA) because no participants were assigned to the arms/groups. Instead, pharmacies from the selected community in each province were assigned to each arm/group (intervention communities and non-intervention communities) rather than participants.
Measure: Number; unit: Number of vaccines administered
Units Other Than Participants: Pharmacies
Arm/Group | Intervention Communities | Non-Intervention Communities
Number analyzed (Participants) | NA | NA
Number analyzed (Pharmacies) | 23 | 21
Number of vaccines administered
  Number of vaccines administered before the intervention (from September 2015 to August 2017) | 3,093 | 5,011
  Number of vaccines administered during the intervention (September 2017 to November 2019) | 6,149 | 5,922

2. Secondary Outcome: Compare the Number of Flu Vaccine Recipients Who Were Recruited and Completed the Online AEFI Survey Among Intervention Pharmacies Using Active Recruitment Strategies and the Non-intervention Pharmacies Using Passive Recruitment Strategies.
Description: Recipients of a flu vaccine in the intervention communities were actively recruited to participate in the CANVAS survey by the intervention pharmacists who handed out information sheets and/or pointed to the QR code to sign up for the survey, while flu vaccine recipients in the non-intervention pharmacies were passively recruited through posters with the QR code displayed in waiting areas without telling them about the study. Note: For this secondary outcome, "recruited" means anyone who signed up for the survey but may not have necessarily completed the survey. The number of flu vaccine recipients who were actively recruited in the intervention pharmacies or passively recruited in the non-intervention pharmacies were compared to assess the effectiveness of the active versus passive recruitment approach.
Time Frame: At the time of survey recruitment, 1 day over the 5-month period the surveys remained open during the influenza seasons
Population: Participants are flu vaccine recipients from both the intervention and non-intervention communities recruited to participate in the survey. Once flu vaccine recipients signed up for the survey, they then received the consent and link to complete the survey, but it was up to their discretion whether they completed the survey. Results show the overall number who signed up for the survey through the active/passive approach, and then the number who decided to complete the survey from each community.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Communities: One community in each Nova Scotia and New Brunswick served as the intervention site where pharmacists used an active recruitment approach for the online AEFI survey, which involved handing out an information sheet and registration form to patients receiving an influenza vaccine in their pharmacies.
- Non-Intervention Communities: One community in each Nova Scotia and New Brunswick served as the non-intervention site where pharmacists used a passive recruitment approach for the online AEFI survey which involved displaying posters and study information sheets that contained a link for the survey patient self-registration page.
Arm/Group | Intervention Communities | Non-Intervention Communities
Number analyzed (Participants) | 365 | 13
Participants | 221 | 8

3. Secondary Outcome: Determining the Awareness About Pharmacists as Immunizers and Vaccination Behaviours of the Targeted Public Using Pre-intervention and Post-intervention Knowledge, Attitudes, Beliefs and Behaviours (KABB) Surveys
Description: As part of the pre- and post-KABB surveys, participants were asked questions regarding their awareness about pharmacists as immunizers and their vaccination behaviour. Questions related to their awareness about pharmacists as immunizers were "Are you aware that many pharmacists are trained to administer vaccines? (Yes or No)" and "Which of the following vaccines are currently administered by pharmacists in a pharmacy? (Check all that apply)". Questions related to their vaccination behaviour were "Did you get or have you ever received... (the following vaccines)?" [Note: Those who answered 'Yes' to these yes/no questions are presented below]
Time Frame: At the time of survey administration, 1 day over the 9-month period each of the surveys remained open
Population: Participants are members of the public from the selected communities who completed the Pre- and Post-Intervention KABB Surveys. They were asked questions about their awareness of pharmacists as immunizers and their vaccination behaviour. There are 3 vaccination behaviour questions that are contingency questions based on the age of the participant and were only asked to those who fall within this age group, which explains why the number analyzed differs from the overall number of participants.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Intervention Knowledge, Attitudes, Beliefs and Behaviours (KABB) Surveys (Public): Before the 2-year demonstration program/intervention (pre-intervention), a cross-sectional online survey was launched to determine the knowledge, attitudes, beliefs, and behaviours (KABB) of community-dwelling adult members of the public. The survey asked questions about the targeted vaccines and the delivery of vaccines by pharmacists and included a variety of yes/no, multiple choice and Likert scale-rating questions.
- Post-Intervention Knowledge, Attitudes, Beliefs & Behaviours (KABB) Surveys (Public): After the 2-year demonstration program/intervention (post-intervention), another cross-sectional online survey was launched to determine the knowledge, attitudes, beliefs, and behaviours (KABB) of community-dwelling adult members of the public regardless of whether or not they were vaccinated as part of this demonstration study. Similar to the pre-intervention survey, this survey asked questions about the targeted vaccines and the delivery of vaccines by pharmacists and included a variety of yes/no, multiple choice and Likert scale-rating questions.
Arm/Group | Pre-Intervention Knowledge, Attitudes, Beliefs and Behaviours (KABB) Surveys (Public) | Post-Intervention Knowledge, Attitudes, Beliefs & Behaviours (KABB) Surveys (Public)
Number analyzed (Participants) | 985 | 992
Participants
  Aware that pharmacists are trained to vaccinate | 850 | 852
  Awareness of pharmacists' ability to administer influenza vaccine | 724 | 680
  Awareness of pharmacists' ability to administer Tdap vaccine | 166 | 122
  Awareness of pharmacists' ability to administer Men ACWY vaccine | 113 | 89
  Awareness of pharmacists' ability to administer MenB vaccine | 113 | 86
  Awareness of pharmacists' ability to administer travel vaccines (hep A, hep B, typhoid vaccines) | NA — This question was not asked to participants during the pre-intervention KABB survey | 327
  Awareness of pharmacists' ability to administer herpes zoster (shingles) | NA — This question was not asked to participants during the pre-intervention KABB survey | 249
  Get the influenza vaccine | 510 | 610
  Ever received Men C or Men ACWY vaccine | 374 | 248
  Ever received Men B vaccine (contingency question for participants between 18-24 years old): number analyzed (Participants) | 364 | 385
  Ever received Men B vaccine (contingency question for participants between 18-24 years old) | 160 | 123
  Ever received Tdap vaccine | 765 | 411
  Ever received high-dose influenza vaccine (contingency question for participants 65 years or older): number analyzed (Participants) | 87 | 86
  Ever received high-dose influenza vaccine (contingency question for participants 65 years or older) | 4 | 12
  Ever received vaccines for travel (hep A, hep B, typhoid vaccines) | NA — This question was not asked to participants during the pre-intervention KABB survey | 530
  Ever received herpes zoster (shingles) vaccine (contingency question for participants 50+): number analyzed (Participants) | 985 | 291
  Ever received herpes zoster (shingles) vaccine (contingency question for participants 50+) | NA — This question was not asked to participants during the pre-intervention KABB survey | 100
  Received all vaccines recommended for adults | 501 | 421
  Ever received a vaccination by a pharmacist in a pharmacy | 384 | 557

4. Secondary Outcome: Determining the Attitudes and Beliefs of the Targeted Public About Pharmacists as Immunizers Using Pre-intervention and Post-intervention Knowledge, Attitudes, Beliefs, and Behaviours (KABB) Surveys
Description: As part of the pre- and post-KABB surveys, participants were asked to indicate how much they agree/disagree with a list of statements about their attitudes and beliefs about pharmacists as immunizers: "Please indicate how much you agree or disagree with the following statements by clicking the box that best fits your opinion". [Note: Those who answered 'agree' are presented below].
Time Frame: At the time of survey administration, 1 day over the 9-month period each of the surveys remained open
Population: Participants are members of the public from the selected communities who completed the Pre- and Post-Intervention KABB Surveys. Participants were asked how much they agree/disagree with a list of statements about their attitudes and beliefs of pharmacists as immunizers [those who answered 'agree' are provided]. In the post-survey, some participants did not respond to the questions, which explains why the number of participants analyzed per row differs from the overall number of participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention Knowledge, Attitudes, Beliefs and Behaviours (KABB) Surveys (Public) | Post-Intervention Knowledge, Attitudes, Beliefs & Behaviours (KABB) Surveys (Public)
Number analyzed (Participants) | 985 | 992
Participants
  I feel comfortable receiving my vaccines from a pharmacist: number analyzed (Participants) | 985 | 896
  I feel comfortable receiving my vaccines from a pharmacist | 739 | 772
  It is convenient for me to receive my vaccines from my pharmacist: number analyzed (Participants) | 985 | 894
  It is convenient for me to receive my vaccines from my pharmacist | 696 | 717
  I think pharmacists have enough training to give vaccines: number analyzed (Participants) | 985 | 896
  I think pharmacists have enough training to give vaccines | 756 | 780
  I would feel more comfortable receiving my vaccines in a pharmacy if my physician recommended it: number analyzed (Participants) | 985 | 896
  I would feel more comfortable receiving my vaccines in a pharmacy if my physician recommended it | 458 | 337
  I would feel more comfortable receiving my vaccines in a pharmacy if a PH nurse recommended it: number analyzed (Participants) | 985 | 896
  I would feel more comfortable receiving my vaccines in a pharmacy if a PH nurse recommended it | 385 | 290
  I would get a vaccine if it was recommended by a doctor: number analyzed (Participants) | 985 | 840
  I would get a vaccine if it was recommended by a doctor | NA — This question was not asked to participants during the pre-intervention KABB survey | 772
  I would get a vaccine if it was recommended by a nurse: number analyzed (Participants) | 985 | 840
  I would get a vaccine if it was recommended by a nurse | NA — This question was not asked to participants during the pre-intervention KABB survey | 738
  I would get a vaccine if it was recommended by a pharmacist: number analyzed (Participants) | 985 | 840
  I would get a vaccine if it was recommended by a pharmacist | NA — This question was not asked to participants during the pre-intervention KABB survey | 692

5. Secondary Outcome: Determining the Awareness of the National Advisory Committee on Immunization (NACI) Guidelines and the Vaccinating Behaviors of Healthcare Providers Through Pre-intervention and Post-intervention Knowledge, Attitudes, Beliefs and Behaviors (KABB) Surveys
Description: As part of the pre- and post-KABB surveys, healthcare providers were asked about their awareness of NACI recommendations and about their vaccinating behaviour. The questions for their awareness of NACI recommendations were "Are you aware that the Canadian guidelines (NACI) recommends/indicates (the following vaccines)". The questions about their vaccinating behaviour was "Do you offer/discuss/recommend (the following vaccines) according to NACI guidelines?" [Note: Those who answered 'Yes' to these yes/no questions are presented below]
Time Frame: At the time of survey administration, 1 day over the 9-month period each of the surveys remained open
Population: Participants are Healthcare Providers (pharmacists, physicians, nurses) in Nova Scotia and New Brunswick who completed the Pre- and Post-Intervention KABB Surveys. Healthcare providers were asked about their awareness of NACI recommendations and their vaccinating behaviour [those who answered 'Yes' are provided]. In the post-survey, some participants did not respond to the questions, which explains why the number of participants analyzed per row differs from the overall number of participants.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Intervention Knowledge, Attitudes, Beliefs and Behaviours (KABB) Surveys (Healthcare Providers): Before the 2-year demonstration program/intervention (pre-intervention), a cross-sectional online survey was launched to determine the knowledge, attitudes, beliefs, and behaviours (KABB) of healthcare providers. The survey asked questions about specific vaccines, current and changing vaccine practices, and logistics of vaccination delivery and included a variety of yes/no, multiple choice, Likert scale-rating questions, and an open-ended question.
- Post-Intervention Knowledge, Attitudes, Beliefs & Behaviours (KABB) Surveys (Healthcare Providers): After the 2-year demonstration program/intervention (post-intervention), another cross-sectional online survey was launched to determine the knowledge, attitudes, beliefs, and behaviours (KABB) of healthcare providers. Similar to the pre-intervention survey, this survey asked questions about specific vaccines, current and changing vaccine practices, and logistics of vaccination delivery and included a variety of yes/no, multiple choice, Likert scale-rating questions, and an open-ended question.
Arm/Group | Pre-Intervention Knowledge, Attitudes, Beliefs and Behaviours (KABB) Surveys (Healthcare Providers) | Post-Intervention Knowledge, Attitudes, Beliefs & Behaviours (KABB) Surveys (Healthcare Providers)
Number analyzed (Participants) | 204 | 223
Participants
  Awareness that NACI recommends that adults receive vaccine for protection against influenza: number analyzed (Participants) | 204 | 173
  Awareness that NACI recommends that adults receive vaccine for protection against influenza | 201 | 163
  Awareness that NACI recommends that older adults (65+) receive a high-dose influenza vaccine: number analyzed (Participants) | 204 | 173
  Awareness that NACI recommends that older adults (65+) receive a high-dose influenza vaccine | 149 | 140
  Awareness that NACI recommends healthy adolescents/young adults receive vaccine for MenACWY: number analyzed (Participants) | 204 | 173
  Awareness that NACI recommends healthy adolescents/young adults receive vaccine for MenACWY | 152 | 133
  Awareness that NACI indicates that healthy adolescents/young adults may receive vaccine for MenB: number analyzed (Participants) | 172 | 138
  Awareness that NACI indicates that healthy adolescents/young adults may receive vaccine for MenB | 112 | 97
  Awareness that NACI recommends that adults receive vaccination for protection against whooping cough: number analyzed (Participants) | 204 | 173
  Awareness that NACI recommends that adults receive vaccination for protection against whooping cough | 163 | 143
  Awareness that CATMAT recommends adults receive travel vaccines depending on where they travel: number analyzed (Participants) | 204 | 173
  Awareness that CATMAT recommends adults receive travel vaccines depending on where they travel | NA — This question was not asked to participants during the pre-intervention KABB survey | 161
  Awareness that NACI recommend that adults 50+ receive a vaccine for protection against shingles: number analyzed (Participants) | 204 | 152
  Awareness that NACI recommend that adults 50+ receive a vaccine for protection against shingles | NA — This question was not asked to participants during the pre-intervention KABB survey | 139
  Discuss the option of receiving the MenB vaccine with eligible adolescents: number analyzed (Participants) | 204 | 148
  Discuss the option of receiving the MenB vaccine with eligible adolescents | 41 | 50
  Recommend that all adolescents who did not get the MenACWY vaccine through school get it: number analyzed (Participants) | 204 | 148
  Recommend that all adolescents who did not get the MenACWY vaccine through school get it | 55 | 66
  Routinely offer all eligible adults the Tdap vaccine: number analyzed (Participants) | 204 | 168
  Routinely offer all eligible adults the Tdap vaccine | 79 | 93
  Offer all eligible adults travel vaccines (Hep A, Hep B, typhoid) according to CATMAT guidelines: number analyzed (Participants) | 204 | 168
  Offer all eligible adults travel vaccines (Hep A, Hep B, typhoid) according to CATMAT guidelines | NA — This question was not asked to participants during the pre-intervention KABB survey | 121
  Offer all eligible adults the shingles vaccines: number analyzed (Participants) | 204 | 168
  Offer all eligible adults the shingles vaccines | NA — This question was not asked to participants during the pre-intervention KABB survey | 132

6. Secondary Outcome: Determining the Attitudes and Beliefs of Healthcare Providers Regarding Pharmacists as Immunizers Using Pre-intervention and Post-intervention Knowledge, Attitudes, Beliefs, and Behaviours (KABB) Surveys
Description: As part of the pre- and post-KABB surveys, healthcare providers were asked about their attitudes and beliefs about pharmacists as immunizers. The questions were: "Where do you think vaccines should be administered? (Check all that apply)" [Note: those who selected 'family doctor's office', 'public health clinic', and/or 'pharmacy' as the locations are presented below]; and "Please indicate how much you agree or disagree with the following statements by clicking the box that best fits your opinion?" [Note: Those who answered 'agree' are presented below].
Time Frame: At the time of survey administration, 1 day over the 9-month period each of the surveys remained open
Population: Participants are Healthcare Providers (pharmacists, physicians, nurses) in Nova Scotia & New Brunswick who completed the Pre- and Post-Intervention KABB Surveys. They were asked about their attitudes and beliefs on pharmacists as immunizers. Some participants did not respond to these questions, which explains why the numbers analyzed differs from the overall numbers of participants. The statement "I would refer a patient to receive a vaccine from a pharmacist" was only asked to physician/nurses.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-Intervention Knowledge, Attitudes, Beliefs and Behaviours (KABB) Surveys (Healthcare Providers) | Post-Intervention Knowledge, Attitudes, Beliefs & Behaviours (KABB) Surveys (Healthcare Providers)
Number analyzed (Participants) | 204 | 223
Participants
  Vaccines should be administered in family doctor's office | 188 | 155
  Vaccines should be administered in public health clinic | 197 | 179
  Vaccines should be administered in pharmacy | 170 | 136
  I support the expansion of pharmacists' scope of practice to include provision of vaccines to adults: number analyzed (Participants) | 204 | 202
  I support the expansion of pharmacists' scope of practice to include provision of vaccines to adults | 171 | 150
  I support the expansion of pharmacist scope of practice to include provision of vaccines to children: number analyzed (Participants) | 204 | 202
  I support the expansion of pharmacist scope of practice to include provision of vaccines to children | 156 | 134
  Pharmacists should be allowed to vaccinate children under the age of 5 years old: number analyzed (Participants) | 204 | 202
  Pharmacists should be allowed to vaccinate children under the age of 5 years old | 66 | 95
  Pharmacists have enough training to administer vaccines: number analyzed (Participants) | 204 | 197
  Pharmacists have enough training to administer vaccines | 136 | 142
  I would refer a patient to receive a vaccine from a pharmacist at a pharmacy (physician/nurses only): number analyzed (Participants) | 83 | 123
  I would refer a patient to receive a vaccine from a pharmacist at a pharmacy (physician/nurses only) | 50 | 75

ADVERSE EVENTS:
Description: All-cause mortality, serious adverse events, and other (not including serious) adverse events were not assessed for the study.
Arm/Group | Intervention Communities | Non-Intervention Communities
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The demonstration program was not able to separate which of the various outreach strategies had the most impact on vaccination uptake (e.g., unable to separate simulated public funding from other outreach strategies such as posters, targeted outreach for the Tdap vaccine). This may be an indication that pharmacies focused on the Tdap vaccine because it was "funded" (simulated public funding).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT02868970/Prot_SAP_000.pdf